CLINICAL TRIAL: NCT06934863
Title: Observational Study of an OLP Patients Cohort: Characteristics, Comorbidities, Risk Factors for Malignant Transformation
Brief Title: Rate of Malignant Transformation and Clinical Characteristics Among an Oral Lichen Planus Cohort: a Retrospective Center Experience
Acronym: LPO_CMR
Status: Recruiting | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Carlo Lajolo, Associate Professor, Catholic University of the Sacred Heart
Other Study IDs: LPO_CMR
Record Dates: First submitted 2025-01-20; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-01

CONDITIONS: Oral Lichen Planus; Oral Carcinoma; Oral Carcinoma in Situ
Keywords: Oral Lichen Planus; Malignant Transformation; Oral Carcinoma; Oral Dysplasia
MeSH Terms: conditions — Lichen Planus, Oral; Mouth Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- A cohort of patients affected by Oral lichen patients: A cohort of patients affected by Oral lichen patients will be evaluated retrospectively in anamnestic and clinical characteristics in order to assess any risk factors for malignant transformation

SUMMARY:
The main objective of this paper will be to evaluate the rate of malignant transformation among a cohort of patients affected by oral lichen planus with long-term follow-up. Secondary aims will be to study and describe the characteristics of these patients to identify potential risk factors for malignant transformation, and to evaluate the therapeutic effects and features to OLP drgus.

DETAILED DESCRIPTION:
Oral Lichen Planus (OLP) is a chronic inflammatory mucocutaneous disease of unknown etiology, primarily affecting the oral mucosa. Global prevalence ranges from 1.01% to 3%, with an estimated 1.43% prevalence in Europe. Although OLP can affect the scalp, nails, and skin, it most commonly manifests in the oral cavity. The disease primarily involves the stratified squamous epithelium of the mouth, and while its precise cause remains unclear, it is thought to result from a T-cell-mediated autoimmune response, triggered by microbial agents, chemicals, stress, or viral infections. T cells directly attack keratinocytes, causing epithelial damage, with both specific (T-cell activity) and nonspecific mechanisms (MMPs, chemokines, and mast cells) contributing to disease progression. CD8+ and CD4+ T cells and Langerhans cells play key roles in antigen presentation, while Matrix Metalloproteinases (MMPs) and their inhibitors (TIMPs) are involved in the breakdown of the basement membrane, leading to keratinocyte destruction.

The main objective of this paper will be to evaluate the rate of malignant transformation among a cohort of patients affected by oral lichen planus with long-term follow-up. Secondary aims will be to study and describe the characteristics of these patients to identify potential risk factors for malignant transformation, and to evaluate the therapeutic effects and features to OLP drgus.

ELIGIBILITY:
Inclusion Criteria:

* Clinical-histological diagnosis of Oral lichen planus
* Patients who gave consensus to personal data treatment
* Minimum 6 months follow-up

Exclusion Criteria:

* Patients who did not give consensus to personal data treatment
* Oral lichenoid lesions
* Patients with anamnesis of hematopoietic stem cells transplant
* Patients with a OSCC at the first histological examination (i.e., namely: also OSCC patients with a OLP background were excluded)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A cohort of patients affected by oral lichen planus
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of Oral Carcinomas | From January 2024 to January 2028
  Number of cases that will be histologically diagnosed as Oral Carcinomas. This outcome will be expressed as a dichotomous variable (i.e., yes/no).

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of the Sacred Heart, Roma, Italy, Italy

IPD SHARING:
Plan to Share IPD: No